CLINICAL TRIAL: NCT06221852
Title: A Randomized Controlled Clinical Trial of Ketogenic and Nutritional Interventions for Brain Energy Metabolism and Psychiatric Symptoms in First Episode Bipolar Disorder.
Brief Title: Ketogenic and Nutritional Interventions for First Episode Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Baszucki Family Foundation (Unknown)
Responsible Party: Principal Investigator, Virginie-Anne Chouinard, MD, Psychiatrist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002849
Record Dates: First submitted 2024-01-11; First posted 2024-01-24 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Bipolar I Disorder; Psychosis; Schizoaffective Disorder
Keywords: First episode psychosis; Ketogenic Diet; Keto; Brain energy metabolism; Insulin resistance; Schizoaffective Disorder; Bipolar Disorder; Magnetic resonance spectroscopy (MRS); Redox; Creatine kinase
MeSH Terms: conditions — Psychotic Disorders; Insulin Resistance; Bipolar Disorder | interventions — Diet, Ketogenic; Nutrition Policy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet arm (Active Comparator): Eligible participants assigned to the ketogenic diet arm will be asked to follow the ketogenic diet (KD) for 12 weeks in addition to any ongoing medications (e.g., mood stabilizers and/or second-generation antipsychotics). Participants will receive weekly and as needed diet counseling from a registered dietician. Participants will be asked to monitor and report their blood ketone levels each day via a finger-prick device provided by the study team. Participants have the ability to opt into an optional open label phase where they can continue on the ketogenic diet with the daily finger pricks for another 12 weeks after the 12-week main study.
  Interventions: Other: Ketogenic diet
- Dietary Guidelines for Americans arm (Active Comparator): Eligible participants assigned to the Dietary Guidelines for Americans (DGA) arm will adhere to the Dietary Guidelines for Americans in addition to any ongoing medications (e.g., mood stabilizers and/or second-generation antipsychotics). Participants will receive weekly and as needed diet counseling from a registered dietician. Participants will be asked to monitor and report their blood ketone levels each day via a finger-prick device provided by the study team. Participants have the ability to opt into an optional open label phase where they can switch to the ketogenic diet with the daily finger pricks for 12 weeks after the 12-week main study.
  Interventions: Other: Dietary Guidelines for Americans

INTERVENTIONS:
Other: Ketogenic diet — The ketogenic diet (KD) is a normo-caloric diet composed of high-fat, low carbohydrate, and adequate protein intake. The KD will consist of 3 meals a day plus snacks, targeting 75-80% fat, 13-18% protein, 7% carbohydrates.
  Arms: Ketogenic diet arm
Other: Dietary Guidelines for Americans — Dietary Guidelines for Americans diet is a normo-caloric diet consisting of 3 meals a day plus snacks, emphasizing nutrient dense foods to meet food group needs (85% of calories), and limits foods and beverages higher in added sugars and saturated fat (15% of calories).
  Arms: Dietary Guidelines for Americans arm

SUMMARY:
This is a randomized, controlled clinical trial to assess the effects of the ketogenic diet in combination with treatment as usual on brain energy metabolism and psychiatric symptoms in individuals with first episode bipolar disorder and schizoaffective disorder.

DETAILED DESCRIPTION:
Several lines of evidence show energy metabolism and redox dysregulation in bipolar disorder and psychotic disorders. Ketogenic interventions targeting energy metabolism are promising therapeutic approaches to improve mood and psychosis in bipolar disorder and other psychotic disorders. Early intervention is also critical to helping people achieve their goals for recovery after a first episode. Investigators aim to use multimodal imaging and metabolic measures to study the effects of a ketogenic diet intervention on energy metabolism and psychiatric symptoms in individuals with first episode bipolar disorder and schizoaffective disorder. This 12-week randomized controlled trial will assess the benefits of a ketogenic diet in combination with treatment as usual compared to a standard diet. Investigators will measure the effects of nutritional ketosis on brain redox and energy metabolism and other neurometabolic markers using magnetic resonance spectroscopy. Furthermore, investigators will measure the effects of the ketogenic diet on mood and psychotic symptoms and metabolic measures such as insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 45.
* Ability to adhere to study diets.
* Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnosis of bipolar I disorder or schizoaffective disorder with onset of illness in the last 7 years.
* Must have a stable psychiatric disorder with no change in psychiatric medications within the past 2 weeks of screening
* Must not be expected to require addition of any new psychiatric medications during the 12-week duration of the study.

Exclusion Criteria:

* Unable to sign informed consent
* Contraindication to magnetic resonance (MR) scan (including claustrophobia)
* Unstable medical illness (including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease)
* Current DSM-5 substance use disorder
* Currently pregnant, nursing, or of childbearing potential and not using a medically accepted means of contraception
* Have a body weight of over 350 lbs or a body mass index (BMI) <20
* Score above 15 on the Young Mania Rating Scale (YMRS)
* History of significant head injury
* Current cancer diagnosis
* Current diagnosis of type 1 or type 2 Diabetes Mellitus
* History of gastric bypass surgery or any weight loss surgery
* Concomitant treatment with Propofol
* Familial hypercholesterolemia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in brain redox nicotinamide adenine dinucleotide metabolites ratio (NAD+/NADH) | 12 weeks
  Change from baseline to week 12 in NAD+/NADH as measured by in vivo phosphorus magnetic resonance spectroscopy (31P-MRS).
Change in brain creatine kinase forward reaction rate (kf) | 12 weeks
  Change from baseline to week 12 in creatine kinase forward reaction rate (kf) as measured by 31P magnetization transfer (MT) MRS.
Change in insulin resistance | 12 weeks
  Change from baseline to week 12 of insulin resistance measured using the homeostatic model assessment of insulin resistance (HOMA-IR) using fasting blood glucose and insulin levels.
Change in psychotic symptoms | 12 weeks
  Change from baseline to week 12 in Positive and Negative Syndrome Scale (PANSS) total score. Scores range from 30-210; a higher score indicates a higher level of psychotic symptoms.
Change in depressive symptoms | 12 weeks
  Change from baseline to week 12 in Hamilton Rating Scale for Depression (HAM-D) total score. Scores range from 0-52; a higher score indicates a higher level of depression.
Change in mania symptoms | 12 weeks
  Change from baseline to week 12 in Young Mania Rating Scale (YMRS) total score. Scores range from 0-60. A higher score indicates a more severe illness.
Change in Clinical Global Impression (CGI) Scale | 12 weeks
  Change from baseline to week 12 in Clinical Global Impression (CGI) Scale. Scores range from 1-7; a higher score indicates higher severity of illness.

SECONDARY OUTCOMES:
Change in body weight | 12 weeks
  Change from baseline to week 12 in participant body weight in kilograms, as measured using a standing scale.
Change in glycated hemoglobin (Hemoglobin A1c) level | 12 weeks
  Change from baseline to week 12 in fasting Hemoglobin A1c level.
Change in triglyceride levels | 12 weeks
  Change from baseline to week 12 in fasting triglyceride levels.
Change in low-density lipoprotein (LDL) levels | 12 weeks
  Change from baseline to week 12 in fasting LDL levels.
Change in high-density lipoprotein (HDL) levels | 12 weeks
  Change from baseline to week 12 in fasting HDL levels.
Change in high-sensitivity C-reactive protein (hs-CRP) levels | 12 weeks
  Change from baseline to week 12 in fasting hs-CRP levels.
Change in brain gamma-aminobutyric acid (GABA) concentration | 12 weeks
  Change from baseline to week 12 in GABA concentration measured by proton magnetic resonance spectroscopy.
Change in brain glutamate metabolite concentration | 12 weeks
  Change from baseline to week 12 in glutamate metabolite concentration measured by proton magnetic resonance spectroscopy.
Change in brain glutathione (GSH) | 12 weeks
  Change from baseline to week 12 in brain GSH measured by proton magnetic resonance spectroscopy.
Change in brain Phosphocreatine (PCr) | 12 weeks
  Changes from baseline to week 12 in PCr concentration as measured by in vivo 31P-MRS.
Change in brain pH | 12 weeks
  Change from baseline to week 12 in pH as measured by in vivo 31P MRS.
Change in brain inorganic phosphate concentration | 12 weeks
  Change from baseline to week 12 in inorganic phosphate (Pi) concentration as measured by in vivo 31P MRS.
Change in adverse events | 12 weeks
  Change from baseline to week 12 from baseline to week 12 in adverse events.
Change in anxiety symptoms | 12 weeks
  Change from baseline to week 12 from baseline to week 12 in Hamilton Anxiety Rating Scale (HAM-A) total score. Scores range from 0 - 56; a higher score indicates a higher level of anxiety.
Change in stress symptoms | 12 weeks
  Change from baseline to week 12 in Depression Anxiety Stress Scales (DASS-42) Stress Subscale score. Scores range from 0-42; a higher score indicates a higher level of stress.
Change in cognitive performance | 12 weeks
  Change from baseline to week 12 in Matrics Consensus Cognitive Battery (MCCB) Total Score. Scores range from 0.00% - 100.00%; a higher score indicates higher cognition.
Change in Global Functioning Scale (GFS) - Social and Role total score | 12 weeks
  Change from baseline to week 12 in Global Functioning Scale (GFS) - Social and Role total score. Scores range from 6-60; a lower score indicates worse social and role functioning.
Change in cell-free mitochondrial DNA (cf-mtDNA) | 12 weeks
  Change from baseline to week 12 in blood and saliva cf-mtDNA levels.
Change in growth differentiation factor 15 (GDF15) | 12 weeks
  Change from baseline to week 12 in blood and saliva GDF15 levels.
Change in blood NAD/NADH+ ratio | 12 weeks
  Change from baseline to week 12 in blood NAD/NADH+ ratio.
Change in blood GSH/GSSH ratio | 12 weeks
  Change from baseline to week 12 in blood GSH/GSSH ratio.

OTHER OUTCOMES:
Change in World Health Organization Disability Assessment Schedule (WHODAS) score | 12 weeks
  Change from baseline to week 12 in World Health Organization Disability Assessment Schedule (WHODAS) scale. Scores range from 0-144. A higher score indicates greater dysfunction and disability in major life domains.
Change in World Health Organization Quality of Life (WHOQOL) score | 12 weeks
  Change from baseline to week 12 in World Health Organization Quality of Life (WHOQOL) scale. Scores range from 1-130. A lower score indicates lower perceived quality of life.
Change in Extrapyramidal Symptom Rating Scale (ESRS) total score | 12 weeks
  Change from baseline to week 12 in Extrapyramidal Symptom Rating Scale (ESRS) total score. Scores range from 0-102; a higher score indicates more severe symptoms.
Change in Pittsburgh Sleep Quality Index (PSQI) total score | 12 weeks
  Change from baseline to week 12 in Pittsburgh Sleep Quality Index (PSQI) total score. Scores range from 0-21; a higher score indicates worse sleep quality.
Change in resting-state fMRI | 12 weeks
  Change within network positive correlations and between network negative correlations from baseline to week 12.
Change in gray matter volume | 12 weeks
  Change in the gray matter volumes (cubic millimeters) of the frontal, parietal and temporal lobes as defined by Freesurfer's Desikan-Killiany Brain Atlas from baseline to week 12.
Change in cortical surface area | 12 weeks
  Change in the cortical surface area (millimeters squared) of the frontal, parietal and temporal lobes as defined by Freesurfer's Desikan-Killiany Brain Atlas from baseline to week 12.
Change in white matter fractional anisotropy (FA) | 12 weeks
  Change in fractional anisotropy (FA), a scalar measure of diffusivity, of water in the brain assessed by DTI at 3T from baseline to week 12. FA values range from 0 (isotropic, meaning diffusion is equally restricted in 3D space) to 1 (anisotrophic, meaning that diffusion is completely restricted to a single direction).

CONTACTS AND LOCATIONS:
Overall Officials: Virginie-Anne Chouinard, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States